CLINICAL TRIAL: NCT02657941
Title: Early and Short Psycho-educational Lifestyle Intervention to Prevent Weight Gain Induced by Psychotropic Drugs in Adults With Severe Mental Illness: a Randomized Controlled Trial
Brief Title: Early and Short Psycho-educational Lifestyle Intervention
Acronym: HYVIE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inclusion problem
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-A00142-47
Record Dates: First submitted 2016-01-13; First posted 2016-01-18 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Obesity; Metabolic Syndrome
MeSH Terms: conditions — Schizophrenia; Obesity; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational group (Experimental): psycho-education program inspired by motivational interviewing and behavioral psychotherapy
  Interventions: Behavioral: Motivational group
- educational group (Active Comparator): exclusively informative psycho-education program
  Interventions: Behavioral: educational group

INTERVENTIONS:
Behavioral: Motivational group — Three weekly sessions of one hour, co-managed by two nurses specialized in psycho-education
  Session 1: General information on the risk of weight gain and the means of prevention, motivational balance on the practice of physical activity, developing a personal goal, information about the sports center Session 2: brainstorming and card game on Food Hygiene Session 3: Find situations at risk of snacking and consider alternative lines
  Arms: Motivational group
Behavioral: educational group — Three weekly sessions of one hour, co-managed by two nurses specialized in psycho-education
  Session 1: General information on the risk of weight gain and means of prevention, video on physical activity, discussions with therapists, information about the sports center Session 2: Video on Food Hygiene, discussions with therapists Session 3: Return on basic concepts covered in the first 2 sessions
  Arms: educational group

SUMMARY:
People with severe mental illness have an increased risk of somatic comorbidities such as metabolic syndrome, obesity, hypertension, dyslipidemia and diabetes mellitus, which induce an increased risk of early mortality, mainly because of cardiovascular diseases.

These high cardio-metabolic risks result of several factors such as lack of access to medical care, a poor and unbalanced nutrition, physical inactivity and smoking but they are also exacerbated by antipsychotic medications and anti-epileptic mood stabilizers prescribed to treat their psychiatric disorder.

These prevention and awareness interventions in lifestyle are most often implemented in ambulatory stabilized patients. Also weight gain occurs in the early months of treatment. The therapeutic education program evaluated in this study seeks to potentiate the effectiveness of these preventive measures through early awareness in hospitalized patients.

Finally, this study aims to compare the efficacy of two early and short programs on health behavior: first a program inspired by motivational interviewing and behavioral psychotherapy and secondly an exclusively educational program (information, formative assessment).

DETAILED DESCRIPTION:
This both psychoeducational programs have a common objective through different methods to promote early awareness of the lifestyle (physical activity and dietary balance) of hospitalized adult patients who receive a psychotropic medication that may cause increased morbidity cardiovascular mortality through excessive weight gain and development of metabolic syndrome.

Both programs have the same number of sessions of the same duration (three weekly sessions of one hour); the same themes are addressed (risk of weight gain and cardiovascular risks induced by treatments, benefits of physical activity and of a balanced diet); only the psycho-educational methods differ.

These programs are for patients with serious mental illness (mainly psychotic disorders and mood disorders), hospitalized in one of the four adult psychiatric units of the Eastern Sector of the Vinatier Hospital in Bron, France. Patients are treatment-naive or already under psychotropic drug(s) but a new antipsychotic or mood-stabilizer must have been started during this hospitalization.

Patients are included on indication of their referring physician in hospital, as soon as their clinical status is compatible. They are randomized to one of two therapeutic educational groups. The two parallel modules of psycho-education are co-managed by two nurses specialized in psycho-education. The study is based on a module per month for 18 months. Patients included will receive three individual interviews with a nurse or psychiatrist: the first interview before module, the second after module and the third three months after module.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients in one of four adult psychiatric units of eastern pole of the Hospital Vinatier
* man or woman
* aged between 18 (major) and 45 years (age limit on inducing a cardiovascular risk)
* receiving anti-psychotic medication or antiepileptic mood stabilizer introduced during this hospitalization: patients must be treatment-naive or already under psychotropic drug(s) since less than 10 years

Exclusion Criteria:

* minor
* aged over 45 years at inclusion
* pregnancy or breastfeeding
* patient suffering from a neurodegenerative disease
* patient suffering from an eating disorder
* patient with a BMI> 30
* patient treated for more than 10 years by anti-psychotic medication or antiepileptic mood stabilizer

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
Change in body weight (kg) | Change from baseline after 3 months

SECONDARY OUTCOMES:
Changes in waist circumference (cm) | Change from baseline after 3 months
  waist circumference measurement during individual interviews standardized assessment (medical or nursing)
Appearance of a SBP (systolic blood pressure) greater than the pathological threshold (> 140 mmHg) or DBP (diastolic blood pressure) above the pathological level (> 90 mmHg) | Change from baseline after 3 months
Appearance of HDL cholesterol below the pathological threshold (<0.40 g/l) and / or LDL cholesterol greater than the pathological threshold (> 2.20 g/l) and / or higher triglyceride pathological level (> 1.5 g/l) | Change from baseline after 3 months
Appearance of a fasting blood glucose higher than pathological threshold defined by ANAES in 1999 (> 1.26 g/l on two samples) | Change from baseline after 3 months
Increased motivation to participate in a non-hospital treatment group on food and cooking | Change from baseline after 3 months
  subjective criterion (declarative) rated on a visual scale in individual interviews standardized assessment (medical or nursing)
Increased motivation to participate in a non-hospital treatment group on physical activity or sport | Change from baseline after 3 months
  subjective criterion (declarative) rated on a visual scale in individual interviews standardized assessment (medical or nursing)
Improved knowledge of balance and food hygiene | Change from baseline after 3 months
  increase of at least 3 points out of 19 in the note obtained during the evaluation done in individual interviews standardized assessment (medical or nursing)

CONTACTS AND LOCATIONS:
Overall Officials: MAGES NICOLAS, PH, Principal Investigator — Responsable de service G08 - Villeurbanne et de l'Unité Polaire de Psychoéducation, Pôle Est, Centre Hospitalier Le Vinatier
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No